CLINICAL TRIAL: NCT04654754
Title: Aerosol Particle Concentrations Among Different Oxygen Devices for Spontaneous Breathing Patients With Tracheostomy: a Randomized Cross-over Trial
Brief Title: Aerosol Particle Concentrations Among Different Oxygen Devices for Spontaneous Breathing Patients With Tracheostomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jie Li (Other)
Responsible Party: Sponsor-Investigator, Jie Li, Associate professor, Rush University Medical Center
Organization: Rush University Medical Center (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: HFOT-trach-aerosol
Record Dates: First submitted 2020-11-25; First posted 2020-12-04 (Actual); Results first posted 2022-11-22 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-11

CONDITIONS: Transmission, Patient-Professional
Keywords: aerosol generating procedure; tracheostomy; oxygen therapy

STUDY DESIGN:
Intervention Model Description: five oxygen and humidification different devices will be used for the enrolled patients, with 5 minutes each. Aerosol particle concentrations at 1 foot away from the patients will be measured.
Who Masked: Outcomes Assessor
Masking Description: the device utilized in the study will be labeled as 1,2,3,4 and 5, the investigator who performed the statistical analysis will be blinded for the device
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (5):
- high-flow high humidity oxygen device with tracheostomy adapter (Experimental): This device provides high-flow gas to tracheostomy patients with heat and humidification. A special adapter is used to connect the tracheostomy tube and circuit.
  Interventions: Device: high-flow high humidity oxygen device with tracheostomy adapter
- large-volume nebulizer (cool aerosol) with trach collar (Active Comparator): This device is the conventional device that is commonly utilized to provide humidification for spontaneous breathing patients with tracheostomy.
  Interventions: Device: high-flow high humidity oxygen device with tracheostomy adapter
- Venturi-adapter with trach collar (Placebo Comparator): This device did not provide any humidification but only oxygen
  Interventions: Device: high-flow high humidity oxygen device with tracheostomy adapter
- large-volume nebulizer (cool aerosol) with T-piece and a filter (Experimental): this device is added with a filter, in order to reduce aerosol particle concentrations in the surrounding environment
  Interventions: Device: high-flow high humidity oxygen device with tracheostomy adapter
- high-flow high humidity device with a scavenger or a surgical mask (Experimental): this device is added with a scavenger or a surgical mask over the adapter, in order to reduce aerosol particle concentrations in the surrounding environment
  Interventions: Device: high-flow high humidity oxygen device with tracheostomy adapter

INTERVENTIONS:
Device: high-flow high humidity oxygen device with tracheostomy adapter — This device can provide heat and humidified gas for spontaneous breathing patients with tracheostomy at a high gas flow rate.
  Other Names: Airvo2, Fisher & Paykel Healthcare Ltd

SUMMARY:
For spontaneous breathing patients with tracheostomy, whose lower airway is directly opened to the room air, the aerosol particles generated by the patients would be directly dispersed into the room air, which might be an direct resource of virus transmission. However, the transmission risk has not been evaluated and the appropriate humidification therapy is unknown. Thus this study is aimed to investigate the aerosol particle concentrations among different oxygen devices for spontaneous breathing patients with tracheostomy, in order to reflect the transmission risk.

DETAILED DESCRIPTION:
The transmission route of the SARS-CoV-2 virus remains controversial, and concerns persist of potentially increased virus transmission when utilizing high-flow devices and aerosol devices among COVID-19 patients. For spontaneous breathing patients with tracheostomy, whose lower airway is directly opened to the room air, the aerosol particles generated by the patients would be directly dispersed into the room air, which might be an direct resource of virus transmission. However, the transmission risk of tracheostomy during spontaneous breathing has not been evaluated and the appropriate humidification therapy is unknown. Thus this study is aimed to investigate the aerosol particle concentrations among different oxygen devices for spontaneous breathing patients with tracheostomy, in order to reflect the transmission risk.

ELIGIBILITY:
Inclusion Criteria:

* adults;
* tracheostomy;
* able to spontaneous breathing without ventilator support

Exclusion Criteria:

* confirmed diagnosis of COVID-19 within recent two weeks;
* non-English speaking;
* refuse to participate in the study;
* palliative care;
* receiving ECMO;
* unable to connect with tracheostomy adapter, such as laryngectomy tube

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-12-23 (Actual); Primary Completion 2021-07-16 (Actual); Study Completion 2021-07-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jie Li, PhD, Principal Investigator — Rush University
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
Data are available upon reasonable request. Proposals should be directed to the corresponding author

REFERENCES:
- [Background] Kaur R, Weiss TT, Perez A, Fink JB, Chen R, Luo F, Liang Z, Mirza S, Li J. Practical strategies to reduce nosocomial transmission to healthcare professionals providing respiratory care to patients with COVID-19. Crit Care. 2020 Sep 23;24(1):571. doi: 10.1186/s13054-020-03231-8. PMID 32967700
- [Result] Dhand R, Li J. Coughs and Sneezes: Their Role in Transmission of Respiratory Viral Infections, Including SARS-CoV-2. Am J Respir Crit Care Med. 2020 Sep 1;202(5):651-659. doi: 10.1164/rccm.202004-1263PP. No abstract available. PMID 32543913
- [Result] Li J, Fink JB, Ehrmann S. High-flow nasal cannula for COVID-19 patients: low risk of bio-aerosol dispersion. Eur Respir J. 2020 May 14;55(5):2000892. doi: 10.1183/13993003.00892-2020. Print 2020 May. PMID 32299867
- [Result] Hui DS, Chow BK, Lo T, Tsang OTY, Ko FW, Ng SS, Gin T, Chan MTV. Exhaled air dispersion during high-flow nasal cannula therapy versus CPAP via different masks. Eur Respir J. 2019 Apr 11;53(4):1802339. doi: 10.1183/13993003.02339-2018. Print 2019 Apr. PMID 30705129
- [Result] Fink JB, Ehrmann S, Li J, Dailey P, McKiernan P, Darquenne C, Martin AR, Rothen-Rutishauser B, Kuehl PJ, Haussermann S, MacLoughlin R, Smaldone GC, Muellinger B, Corcoran TE, Dhand R. Reducing Aerosol-Related Risk of Transmission in the Era of COVID-19: An Interim Guidance Endorsed by the International Society of Aerosols in Medicine. J Aerosol Med Pulm Drug Deliv. 2020 Dec;33(6):300-304. doi: 10.1089/jamp.2020.1615. Epub 2020 Aug 12. PMID 32783675
- [Result] Rovira A, Dawson D, Walker A, Tornari C, Dinham A, Foden N, Surda P, Archer S, Lonsdale D, Ball J, Ofo E, Karagama Y, Odutoye T, Little S, Simo R, Arora A. Tracheostomy care and decannulation during the COVID-19 pandemic. A multidisciplinary clinical practice guideline. Eur Arch Otorhinolaryngol. 2021 Feb;278(2):313-321. doi: 10.1007/s00405-020-06126-0. Epub 2020 Jun 17. PMID 32556788
- [Result] McGrath BA, Brenner MJ, Warrillow SJ, Pandian V, Arora A, Cameron TS, Anon JM, Hernandez Martinez G, Truog RD, Block SD, Lui GCY, McDonald C, Rassekh CH, Atkins J, Qiang L, Vergez S, Dulguerov P, Zenk J, Antonelli M, Pelosi P, Walsh BK, Ward E, Shang Y, Gasparini S, Donati A, Singer M, Openshaw PJM, Tolley N, Markel H, Feller-Kopman DJ. Tracheostomy in the COVID-19 era: global and multidisciplinary guidance. Lancet Respir Med. 2020 Jul;8(7):717-725. doi: 10.1016/S2213-2600(20)30230-7. Epub 2020 May 15. PMID 32422180
- [Result] Birk R, Handel A, Wenzel A, Kramer B, Aderhold C, Hormann K, Stuck BA, Sommer JU. Heated air humidification versus cold air nebulization in newly tracheostomized patients. Head Neck. 2017 Dec;39(12):2481-2487. doi: 10.1002/hed.24917. Epub 2017 Oct 9. PMID 28990261

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is a randomized crossover study, all the 12 patients received the five treatments in a random order.
Groups:
- Spontaneous Breathing Patients With Tracheostomy: Patients who received tracheostomy and had spontaneous breathing, without ventilator support
Period: LVN With T-piece and a Filter
Arm/Group | Spontaneous Breathing Patients With Tracheostomy
Started | 12
Completed | 12
Not Completed | 0
Period: High-flow High-humidity With Adapter
Arm/Group | Spontaneous Breathing Patients With Tracheostomy
Started | 12
Completed | 12
Not Completed | 0
Period: LVN With Trach Collar
Arm/Group | Spontaneous Breathing Patients With Tracheostomy
Started | 12
Completed | 12
Not Completed | 0
Period: Venturi With Trach Collar
Arm/Group | Spontaneous Breathing Patients With Tracheostomy
Started | 12
Completed | 12
Not Completed | 0
Period: High-flow High-humidity With Scavenger
Arm/Group | Spontaneous Breathing Patients With Tracheostomy
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Spontaneous Breathing Patients With Tracheostomy: Patients who had tracheostomy and spontaneous breathing, without ventilator support
Arm/Group | Spontaneous Breathing Patients With Tracheostomy
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.5 (16.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Aerosol Particle Concentrations With Size of 1-3 Micrometer at 1 Foot Away From the Patient
Description: aerosol particle concentrations (the concentrations of particles inside the room air, the unit is particles per cubic meters) at 1 foot away from the patient
Time Frame: 5 minutes after using the device
Measure: Median (Inter-Quartile Range); unit: particles/m3
Groups:
- Spontaneous Breathing Patients With Tracheostomy: Patients who had tracheostomy and could breathe spontaneously without ventilator support
Arm/Group | Spontaneous Breathing Patients With Tracheostomy
Number analyzed (Participants) | 12
particles/m3
  High-flow High Humidity Oxygen Device With Tracheostomy Adapter | 13000 [10000 to 31000]
  Large-volume Nebulizer (Cool Aerosol) With Trach Collar | 11000 [6000 to 29000]
  Venturi-adapter With Trach Collar | 10000 [8000 to 23000]
  Large-volume Nebulizer (Cool Aerosol) With T-piece and a Filter | 12000 [7000 to 26000]
  High-flow High Humidity Device With a Scavenger or a Surgical Mask | 13000 [9000 to 25000]

2. Primary Outcome: Aerosol Particle Concentrations With Size of <0.3 Micrometer at 1 Foot Away From the Patient
Description: as for outcome 1
Time Frame: 5 minutes after using the device
Measure: Median (Inter-Quartile Range); unit: particles/m3
Arm/Group | Spontaneous Breathing Patients With Tracheostomy
Number analyzed (Participants) | 12
particles/m3
  High-flow High Humidity Oxygen Device With Tracheostomy Adapter | 10500000 [7700000 to 23000000]
  Large-volume Nebulizer (Cool Aerosol) With Trach Collar | 15200000 [7200000 to 26000000]
  Venturi-adapter With Trach Collar | 12100000 [6900000 to 26600000]
  Large-volume Nebulizer (Cool Aerosol) With T-piece and a Filter | 11900000 [7300000 to 25500000]
  High-flow High Humidity Device With a Scavenger or a Surgical Mask | 13000000 [7900000 to 25400000]

3. Primary Outcome: Aerosol Particle Concentrations With Size of 0.3-0.5 Micrometer at 1 Foot Away From the Patient
Description: as for outcome 1
Time Frame: 5 minutes after using the device
Measure: Median (Inter-Quartile Range); unit: particles/m3
Arm/Group | Spontaneous Breathing Patients With Tracheostomy
Number analyzed (Participants) | 12
particles/m3
  High-flow High Humidity Oxygen Device With Tracheostomy Adapter | 610000 [460000 to 1790000]
  Large-volume Nebulizer (Cool Aerosol) With Trach Collar | 730000 [380000 to 3150000]
  Venturi-adapter With Trach Collar | 610000 [360000 to 1210000]
  Large-volume Nebulizer (Cool Aerosol) With T-piece and a Filter | 590000 [390000 to 1760000]
  High-flow High Humidity Device With a Scavenger or a Surgical Mask | 680000 [410000 to 1960000]

4. Primary Outcome: Aerosol Particle Concentrations With Size of 0.5-1 Micrometer at 1 Foot Away From the Patient
Description: as for outcome 1
Time Frame: 5 minutes after using the device
Measure: Median (Inter-Quartile Range); unit: particles/m3
Arm/Group | Spontaneous Breathing Patients With Tracheostomy
Number analyzed (Participants) | 12
particles/m3
  High-flow High Humidity Oxygen Device With Tracheostomy Adapter | 53000 [35000 to 137000]
  Large-volume Nebulizer (Cool Aerosol) With Trach Collar | 55000 [36000 to 140000]
  Venturi-adapter With Trach Collar | 46000 [36000 to 132000]
  Large-volume Nebulizer (Cool Aerosol) With T-piece and a Filter | 52000 [36000 to 101000]
  High-flow High Humidity Device With a Scavenger or a Surgical Mask | 50000 [42000 to 139000]

5. Primary Outcome: Aerosol Particle Concentrations With Size of 3-5 Micrometer at 1 Foot Away From the Patient
Description: as for outcome 1
Time Frame: 5 minutes after using the device
Measure: Median (Inter-Quartile Range); unit: particles/m3
Arm/Group | Spontaneous Breathing Patients With Tracheostomy
Number analyzed (Participants) | 12
particles/m3
  High-flow High Humidity Oxygen Device With Tracheostomy Adapter | 6700 [5300 to 15200]
  Large-volume Nebulizer (Cool Aerosol) With Trach Collar | 6000 [2500 to 15500]
  Venturi-adapter With Trach Collar | 5700 [4600 to 12000]
  Large-volume Nebulizer (Cool Aerosol) With T-piece and a Filter | 6000 [3500 to 14100]
  High-flow High Humidity Device With a Scavenger or a Surgical Mask | 6700 [4900 to 12700]

6. Primary Outcome: Aerosol Particle Concentrations With Size of 5-10 Micrometer at 1 Foot Away From the Patient
Description: as for outcome 1
Time Frame: 5 minutes after using the device
Measure: Median (Inter-Quartile Range); unit: particles/m3
Arm/Group | Spontaneous Breathing Patients With Tracheostomy
Number analyzed (Participants) | 12
particles/m3
  High-flow High Humidity Oxygen Device With Tracheostomy Adapter | 3500 [2100 to 7100]
  Large-volume Nebulizer (Cool Aerosol) With Trach Collar | 3200 [1400 to 7400]
  Venturi-adapter With Trach Collar | 3900 [1800 to 4600]
  Large-volume Nebulizer (Cool Aerosol) With T-piece and a Filter | 3500 [2500 to 6400]
  High-flow High Humidity Device With a Scavenger or a Surgical Mask | 3200 [2500 to 5300]

7. Secondary Outcome: Patient Comfort With Different Oxygen Devices
Description: Patients would scale their comfort on a 5-point Likert scale, 1 was the most uncomfortable, and 5 was the most comfortable.
Time Frame: 5 minutes after using the device
Measure: Mean (Standard Deviation); unit: score on a scale (comfort scores 1-5)
Arm/Group | Spontaneous Breathing Patients With Tracheostomy
Number analyzed (Participants) | 12
score on a scale (comfort scores 1-5)
  High-flow High Humidity Oxygen Device With Tracheostomy Adapter | 3.5 (1.5)
  Large-volume Nebulizer (Cool Aerosol) With Trach Collar | 3.8 (1.3)
  Venturi-adapter With Trach Collar | 3.5 (1.2)
  Large-volume Nebulizer (Cool Aerosol) With T-piece and a Filter | 3.3 (1.3)
  High-flow High Humidity Device With a Scavenger or a Surgical Mask | 3.5 (1.2)

ADVERSE EVENTS:
Time Frame: 3 hours
Arm/Group | Spontaneous Breathing Patients With Tracheostomy
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-12-13): https://cdn.clinicaltrials.gov/large-docs/54/NCT04654754/Prot_SAP_000.pdf
  • Informed Consent Form (2020-12-13): https://cdn.clinicaltrials.gov/large-docs/54/NCT04654754/ICF_001.pdf